CLINICAL TRIAL: NCT02885792
Title: Coronary Artery Disease as a Cause of Morbidity and Mortality in Patients Suffering From Schizophrenia: Epidemiology and Status to Provide Prevention, Interventions and Treatment
Brief Title: Coronary Artery Disease in Patients Suffering From Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg Psychiatric Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Aagaard, Chief consultant, Professor, Dr.Med.Sci., Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N-20140047
Record Dates: First submitted 2016-07-01; First posted 2016-09-01 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Schizophrenia; Cardiovascular Disease
Keywords: Schizophrenia; Cardiovascular disease; Premature mortality; Arteriosclerosis; Risk factor; Intervention; Treatment; Somatic morbidity
MeSH Terms: conditions — Schizophrenia; Cardiovascular Diseases; Arteriosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Debuting and chronic schizophrenia (Experimental): ILLNESS HISTORY:
  * Existing psychiatric and somatic diagnosis and treatment
  * Charlson co-morbidity
  MEASURE OF SOCIAL CONDITIONS
  - For example Lubben Social Network Scale-6 and Brief Trauma Questionnaire.
  MEASURE OF PSYCHIATRIC CONDITION::
  * Positive and Negative Syndrome Scale (PANSS)
  * Clinical Global Impression Scale (CGI)
  * Columbia Suicide Severity Rating Scale (C-SSRS)
  * Beck Cognitive Insight Scale
  * Birchwood Insight Scale
  CARDIOVASCULAR MEASUREMENT:
  CT Coronary angiography (CT-CAG)
  * Echocardiography
  * Heart rate variability (HRV)
  * Pulmonary function test (PFT)
  * Toe blood pressure (TBP)
  * Blood test
  * Body composition analysis
  * CT scan of upper abdomen
  * Cardiovascular magnetic resonance imaging (CMR)
  * Adipose tissue biopsy
  Interventions: Other: Illness history; Other: Measure of social conditions; Other: Measure of psychiatric condition; Procedure: Cardiovascular measurement
- Matched controls (Active Comparator): CARDIOVASCULAR MEASUREMENT:
  * CT Coronary angiography (CT-CAG)
  * Echocardiography
  * Heart rate variability (HRV)
  * Pulmonary function test (PFT)
  * Toe blood pressure (TBP)
  * Blood test
  * Body composition analysis
  * CT scan of upper abdomen
  * Cardiovascular magnetic resonance imaging (CMR)
  * Adipose tissue biopsy
  Interventions: Procedure: Cardiovascular measurement

INTERVENTIONS:
Other: Illness history — Existing psychiatric and somatic diagnosis and treatment. Charlson co-morbidity Index.
  Arms: Debuting and chronic schizophrenia
Other: Measure of social conditions — A self-report questionnaire measuring social isolation, including relations to family and friends.
  Arms: Debuting and chronic schizophrenia
Other: Measure of psychiatric condition — This method measures symptom severity, therapeutic response and general improvement, suicidal ideation, cognitive insight and awareness of illness and need for treatment and the ability to relabel symptoms.
  Arms: Debuting and chronic schizophrenia
Procedure: Cardiovascular measurement — This procedure is used to detect early identification of cardiovascular disease progression.

SUMMARY:
Schizophrenia is a severe mental illness associated with excess mortality and affecting nearly 1% of the population. The average life expectancy for patients diagnosed with schizophrenia has been 55-60 years through the last generations in Denmark, while the general population has over the same period of time experienced an increase in life expectancy. As a result, the standardized mortality rate for patients with schizophrenia has increased markedly over the last three decades and is currently a major public health concern. Causes of death are mainly cardiovascular disease and patients diagnosed with schizophrenia has a relative risk of cardiovascular disease that is about 2-fold higher than the general population.

DETAILED DESCRIPTION:
Little is known about severe progression of premature coronary arteriosclerosis in patients suffering from schizophrenia. Coronary artery calcium score is a well-defined measure to predict cardiovascular disease events, however there has not yet been any attempt to investigate whether there is an association between coronary artery calcium score and premature morbidity and mortality in patients diagnosed with schizophrenia.

The objective of this study is to investigate the progression of arteriosclerosis in patients with schizophrenia at different stages of the disease, and to offer and implement adequate treatment for these patients according to their somatic condition. This study will identify risk factors of somatic diseases in these patients, with specific focus on early diagnoses, prevention, intervention and treatment of arteriosclerosis in schizophrenic patients.

The investigation is about the possibility of detecting any differences between developing arteriosclerosis in schizophrenia patients versus the general population, and how common risk factors are contributing to this process. The results of this study should provide important modifications in the clinical guidelines for treatment of patients diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of F20 schizophrenia.
* Informed statement of consent
* Age > 18

Exclusion Criteria:

* Incompetency to create stabile relation or make agreements
* Pregnancy and also breastfeeding women
* Participants with severe claustrophobia
* Participants with lack of ability to cooperate with the planned study program.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
CT coronary angiography - a quantitative clinical measurement | 6 years
  CT coronary angiography is a non-invasive procedure that uses simple CT-scan without contrast to measure coronary calcifications

SECONDARY OUTCOMES:
Existing psychiatric and somatic diagnosis and treatment - Self-report questionnaire | 6 years
  Measure of illness history with focus on previous diagnosis and treatment
Charlson Co-morbidity index - Self-report questionnaire | 6 years
  Measure of illness history with focus on which additional somatic or psychiatric diagnosis patients have.
Lubben Social Network Scale-6 (LSNS-6) - Self-report questionnaire | 6 years
  The LSNS-6 is a self-report questionnaire measuring social isolation, including relations to family and friends.
Global Assessment of Functioning (GAF) - Clinical evaluation | 6 years
  The GAF is a clinical evaluation of the patient's overall functioning level, including psychological, social and interpersonal, and occupational functioning of mental health-illness.
Positive and Negative Syndrome Scale (PANNS) - Clinical psychiatric evaluation | 6 years
  The PANNS measures symptom severity in schizophrenia with focus on two distinct syndromes. The postive syndromes including productive symptoms, and the negative syndrome, including deficit features.
Clinical Global Impression Scale (CGI) - Clinical psychiatric evaluation | 6 years
  The CGI is a measure of symptom severity, therapeutic response and general improvement.
Echocardiography - Clinical objective evaluation | 6 years
  Echocardiography is a non-invasive procedure that uses ultrasound waves to generate live images of the patient's heart
Heart rate variability (HRV) - Clinical objective evaluation | 6 years
  HRV is a non-invasive procedure that detects the function of the autonomic nervous system on the heart rhythm.
Pulmonary function test (PFT) - Clinical objective evaluation | 6 years
  PFT also known as spirometry is a procedure that measures lung function
Toe brachial index (TBI) - Clinical objective evaluation | 6 years
  TBP is a procedure that measures the relationship between the systolic blood pressure at the toe and the arm
Blood test - Clinical objective evaluation | 6 years
  Blood test is used to identify biomedical markers. A volume of 20 ml will be needed from each patient.
Body Composition analysis (BCA) - Clinical objective evaluation | 6 years
  Using a standard weight to measure body composition for each patient
CT-scan of upper abdomen (CTUA) - Clinical objective evaluation | 6 years
  CTUA uses X-rays to produce cross-sectional images of the heart and liver
Cardiovascular magnetic resonance imaging(CMR) - Clinical objective evaluation | 6 years
  CMR uses a strong magnetic field including radio waves to generate images of the heart
Adipose tissue biopsy - Clinical objective evaluation | 6 years
  Adipose tissue biopsy is an invasive procedure that we use to understand the composition of fat acid for each patient in order to understand the correlation between fat acid and cardiovascular disease.
Urine sample - Objective clinical evaluation | 6 years
  Urine sample measures the content of melatonin, which is a hormone that controls the natural cycle of sleeping and waking hours.

CONTACTS AND LOCATIONS:
Overall Officials: Svend E. Jensen, MD, Principal Investigator — Aalborg University Hospital, Psychiatric Hospital
Locations (1):
- Aalborg University Hospital, Psychiatric Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jorgensen LR, Hegtmann CL, Straszek SPV, Hoyer C, Polcwiartek C, Petersen LJ, Dalgaard MK, Jensen SE, Nielsen RE. Peripheral artery disease in patients with schizophrenia as compared to controls. BMC Cardiovasc Disord. 2023 Mar 8;23(1):126. doi: 10.1186/s12872-023-03143-9. PMID 36890440
- [Derived] Trab T, Attar R, Jensen SE, Grontved S, Frokjaer JB, Polcwiartek C, Nielsen RE. Coronary artery calcium in patients with schizophrenia. BMC Psychiatry. 2021 Aug 23;21(1):422. doi: 10.1186/s12888-021-03412-x. PMID 34425769